CLINICAL TRIAL: NCT00215319
Title: A Multi-center Study to Evaluate the Safety and Efficacy of DePuy AcroMed Titanium Surgical Mesh and MOSS-Miami Spinal Fixation System Pedicle Screws for Intradiscal Fusion in the Lumbar Spine
Brief Title: Titanium Surgical Mesh and MOSS-Miami Screws for Lumbar Fusion.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G990313
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative disc disease at up to 2 levels (L2-S1)
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Pedicle Screws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TSM Cage (Experimental): Lumbar I/F with cage and pedicle screws
  Interventions: Device: Lumbar I/F with cage and pedicle screws

INTERVENTIONS:
Device: Lumbar I/F with cage and pedicle screws — Surgical Titanium Mesh™ with MOSS-Miami™ Pedicle Screws

SUMMARY:
The purpose of this study is to determine the clinical success of DePuy Spine Titanium Surgical Mesh with MOSS Miami Spinal Fixation System Pedicle Screws in the treatment of one or two levels of degenerative disc disease of the lumbar spine. The observed success rate at 24 months will be compared to an historical control group treated with the Lumbar I/F Cage with VSP System.

DETAILED DESCRIPTION:
This is a single arm multi-center study to determine the clinical success of the DePuy Spine Titanium Surgical Mesh with MOSS Miami Spinal Fixation System Pedicle Screws in the treatment of one or two adjacent levels of degenerative disc disease of the lumbar spine (L2 - S1).

Study Success is as a compound endpoint requiring:

* Radiographic Fusion,
* Improvement in Pain/Function,
* Maintenance/Improvement in Neurologic Status, and
* Freedom from Secondary Surgical Intervention.
* The rate of Adverse Events must be no worse than in the control group as well.

Secondary Endpoints Include:

* Adverse Events
* SF-36 Health Related Quality of Life
* Disc Space Height
* Work Status

Comparison:

Results will be compared to an historical control group treated with the Lumbar I/F Cage with VSP System.

ELIGIBILITY:
Inclusion Criteria:

* Persistent back and/or leg pain refractory to 6 months of non-surgical therapy
* Radiographic evidence of significant disc degeneration at one or two of the adjacent lumbar levels L2-S1.

Exclusion Criteria:

* Abnormality at more than two levels,
* Prior fusion surgery of the lumbar spine; prior discectomies or IDET allowed,
* Infection in the disc or spine, past or present,
* Active infection at time of surgery,
* Tumor in the spine,
* Significant osteoporosis or metabolic bone disease,
* Greater than Grade I spondylolisthesis or significant bony defect in the lumbar spine,
* Pregnant or lactating, or wishes to become pregnant within duration of study,

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2000-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Radiographic Fusion
Oswestry Disability Index
Motor Function
Adverse Events
Secondary Surgical Interventions

SECONDARY OUTCOMES:
SF-36
Graft site pain
Back pain
Leg pain
Disc space height

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TSM Investigational Site A, Dothan, Alabama
  - TSM Investigational Site B, Fort Wayne, Indiana